CLINICAL TRIAL: NCT05724004
Title: A-SAB - Alectinib Followed by Concomitant Consolidation SBRT/Hypofractionated Radiation Therapy/SRS in Advanced NSCLC With ALK-rearrangement
Brief Title: Alectinib Followed by Concomitant Consolidation Radiation Therapy in Advanced NSCLC With ALK-rearrangement (A-SAB)
Acronym: A-SAB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Karin Lindberg, Principal investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A-SAB
Record Dates: First submitted 2023-01-20; First posted 2023-02-13 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Radiotherapy Side Effect; Non-small Cell Lung Cancer; ALK Gene Mutation
Keywords: Stereotactic body radiation therapy; SBRT; Radiotherapy; Non-small Cell Lung Cancer; ALK-rearrangement
MeSH Terms: conditions — Radiation Injuries; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: Single arm, multicenter, phase I/II study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy + alectinib (Experimental): All patients receive consolidation radiation therapy to all active tumour lesions after induction treatment with alectinib.
  Interventions: Radiation: SBRT/SRS/radiation therapy

INTERVENTIONS:
Radiation: SBRT/SRS/radiation therapy — Consolidation radiation therapy (SBRT/SRS/moderately hypofractionated radiation therapy)

SUMMARY:
The goal of this clinical trial is to learn evaluate the safety and efficacy of the addition of radiation therapy to all tumour lesions, to first line medical treatment with alectinib in non-small cell lung cancer harbouring ALK-rearrangements.

The main aims of the trial are to evaluate:

* if the treatment combination is safe
* if the treatment combination can inhibit progression

Participants who have responded to 1st line alectinib will be treated with consolidation radiation therapy to all remaining tumour lesions while continuing on alectinib until disease progression, unacceptable toxicity or another discontinuation criterion is met.

DETAILED DESCRIPTION:
This is phase I/II study to evaluate the feasibility (phase I) and progression free survival (phase II) in patients with advanced NSCLC with ALK-rearrangement receiving consolidation radiation therapy (RT) to all known macroscopic tumour lesions present after 2-3 months of treatment with alectinib and then continuing with alectinib.

Eligible patients are those with an ALK-rearranged stage III (non-surgical/non-radiochemotherapy candidates) OR stage IV NSCLC who, after a 2-3-month-induction period of alectinib show stable disease/partial response to systemic therapy. When entering the trial, all known tumour lesions are treated with SBRT/RT/SRS with concomitant alectinib followed by continuation alectinib until disease progression, unacceptable toxicity or another discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological confirmed NSCLC:

   * Stage IV NSCLC OR
   * Stage III NSCLC not suitable for surgery or radiochemotherapy OR
   * Recurrent NSCLC after previous surgery (not amendable for curative multimodal therapy)
2. ALK-rearrangement
3. Adequate organ function to tolerate alectinib and clinical tolerance to alectinib
4. Stable disease (SD) or partial response (PR) after 2-3 months induction treatment with alectinib
5. Maximum 5 tumour lesions +/- thoracic lymph nodes active on an 18F-FDG-PET scan post induction treatment with alectinib
6. All active tumour lesions amendable to RT under the following conditions:

   * All metastases possible to treat with

     * Extracranial metastases: SBRT of at least 7 Gy x 5 (corresponding to 50 Gy EQD2 using alfa/beta 10Gy)
     * Intracranial metastases: SRS or f-SRS
   * The primary tumour and/or lymph nodes and/or pulmonary metastases amendable to SBRT (≥ 7Gy x 5, see above) or moderately hypofractionated RT of 3 Gy x 15 (corresponding to 49 Gy EQD2 using alfa/beta 10Gy)
7. Adequate organ function to tolerate SBRT/RT:

   * Fulfilment of dose constraints to adequate organs at risk
8. ECOG performance status (PS) 0-2
9. FEV1 ≥1 litre (only applicable for lung targets)
10. Age ≥ 20 years
11. Measurable lesions according to RECIST v 1.1
12. Signed written informed consent

Exclusion Criteria:

1. Leptomeningeal carcinosis (on MRI or in cerebrospinal fluid (CSF))
2. Persistent malignant pleural effusion, malignant pericardial effusion or malignant ascites after induction treatment
3. PD after 2-3-month-induction treatment with alectinib
4. Previous TKI, chemotherapy or immunotherapy (previous adjuvant chemotherapy for early stage NSCLC is allowed) for metastatic NSCLC
5. Previous RT for NSCLC (any stage)
6. Previous RT for any other cancer within the last 3 years possibly interfering with the planned RT within this study
7. Life expectancy of less than 6 months
8. Inability to understand given information or undergo study procedures according to protocol.
9. Has evidence or a past medical history of interstitial lung disease or active, non-infectious pneumonitis or known pulmonary fibrosis.
10. Pregnant or breast-feeding. Patients must agree to use safe contraception during and for 3 months after study treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2031-06-20 (Estimated)

PRIMARY OUTCOMES:
Toxicity (safety) | 6 months post radiation therapy
  No and percentage of patients suffering grade 3-5 toxicity attributed to RT and within 6 months post RT).
Progression free survival (PFS) | PFS rate at 12 months after initiation of alectinib
  PFS-rate at 12 months (KM-estimated method). Successrate is 12-month-PFS-rate of 85%. Median PFS will also be measured

SECONDARY OUTCOMES:
Overall survival | 5 years
  OS-rate at 1-, 2-, 3- and 5 years post initiation of alectinib using the KM-method. Median OS will also be measured.
Progression free survival II | 5 years
  (Time between the date of initiation of alectinib and the date of documented 2nd tumour progression or death, from whatever reason.) PFS II rate at 1-, 2-, 3- and 5 years (KM-method) will be measured.
Time to treatment failure | 3 years
  Time between the date of initiation of alectinib and the date of documented progressive disease, unacceptable toxicity related to SBRT, toxicity attributed to alectinib leading to interruption of the treatment or death. (Time between the date of initiation of alectinib and the date of documented 2nd tumour progression or death, from whatever reason.) TTF-rate at 1-, 2-, 3- and 5 years (KM-method).
Time to next therapy | 5 years
  Time between the date of initiation of alectinib and the date of next therapy. (Time between the date of initiation of alectinib and the date of documented 2nd tumour progression or death, from whatever reason.) Rate at 1-, 2-, 3- and 5 years (KM-method).

OTHER OUTCOMES:
Translational biomarker studies | 5 years
  For plasma samples: extracellular vesicles isolated from plasma are profiled for protein and RNA expression with linkage to clinical response and tumor marker expression.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Lindberg, MD, PhD, Study Director — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No